CLINICAL TRIAL: NCT00982215
Title: Pilot Study of Pharmacology of Paracetamol Administered Per-oral Mucosa
Acronym: PMB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Unither Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0057
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Paracetamol; per-oral mucosa PMB; No disease, healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Kinetics of plasma concentrations of paracetamol — Pilot study of Pharmacology Paracetamol administered per-oral mucosa PMB. Crossover study, double-blind, randomized, controlled versus placebo.
Drug: Placebo — Pilot study of Pharmacology Paracetamol administered per-oral mucosa PMB. Crossover study, double-blind, randomized, controlled versus placebo.

SUMMARY:
Paracetamol is the centrally acting analgesic most commonly used in the world, indicated for the symptomatic treatment of fever and pain in mild to moderate. It comes in different formulations for oral, intravenous and rectal. The IV route allows rapid passage of paracetamol in the systemic arterial circulation and thus the brain, faster distribution evidenced a higher plasma concentration compared with oral and rectal. However the IV route also has disadvantages well known risks iatrogenic perfusion is an invasive lengthy, unpleasant and painful.

The way per-Albus not to date used for the administration of paracetamol. It is a path nonetheless very interesting for the rapid absorption of drugs such as nitrates used in angina pectoris, as it seeks a highly vascular area (the floor of the tongue or gingival groove) and allows a very rapid action. Furthermore, the terminal per-oral mucosa, less restrictive than IV administration and faster than oral administration, requires a simple medical gesture without special surveillance after administration, produces no pain or risk of infection for the patient (in contrast to the IV). It is interesting to test a new dosage form per-oral mucosa of paracetamol and compare pharmacological level (pharmacokinetics and pharmacodynamics) with the only dosage form of reference used by the IV route.

DETAILED DESCRIPTION:
Pilot study of Pharmacology Paracetamol administered per-oral mucosa PMB. Crossover study, double-blind, randomized, controlled versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged over 18 years and not more than 50 years
* Males
* Values of vital signs before administration of the test products:

  * NOT between 100-140 mm Hg
  * PAD between 50-90 mm Hg
  * Radial pulse between 45-90 beats per minute
* Free from any treatment in the 7 days preceding inclusion including no use of analgesics or anti-inflammatories)

Exclusion Criteria:

* Contraindications to the administration of paracetamol
* Hypersensitivity to paracetamol
* History of hepatitis B or C
* Severe renal impairment
* Hepatic insufficiency
* Medical history and / or surgical judged by the investigator or his representative as being incompatible with the test, especially subjects with neuropathic pain
* Pathology evolutionary time of the review for inclusion
* Binge drinking, smoking (more than 10 cigarettes/day), coffee, tea or drinks containing caffeine (equivalent to more than 4 cups per day) or drug abuse
* Subject does not meet the selection criteria regarding their ability to discriminate the sensations resulting from noxious stimuli during psychometric testing
* Topic having all breaches of the oral mucosa (aphthae)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Kinetics of plasma concentrations of paracetamol | after administration of paracetamol

SECONDARY OUTCOMES:
Change in pain threshold testing mechanical stimulation (von Frey electronic). Follow-up to the pain assessed by VAS (visual analog rating) | after administration of paracetamol
Variation of the amplitude of brain wave N2P2 induced thermal stimulus at the forearm (Evoked Potentials thermal) | after administration of paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — University Hospital, Clermont-Ferrand